CLINICAL TRIAL: NCT01945463
Title: The Effect of Breast Augmentation on the Quality of Echocardiography Test
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0378-13
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-08

CONDITIONS: Breast Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast augmentation surgery is currently the most common elective plastic surgery performed in the US. With regards to the surgical technique, there are 4 incisional sites available for breast augmentation, each with its advantages and disadvantages: Axillary, Periareolar, inframammary, and umbilical. The implant is inserted in either a subglandular (beneath breast tissue), submuscular (underneath the Pectoralis Major), or "dual-plane" (combination of both) manner.

Echocardiography is the most commonly used diagnostic test in cardiology for the evaluation of cardiac structure and function. Its use has increased dramatically in the last decades. We have encountered three women with congenital heart disease who have undergone breast augmentation, and their echocardiographic images were significantly limited after the implantation. There is only one case report in the medical literature suggesting that breast implants interfere with echocardiographic views .

The underlying physical property of the silicone breast implants that causes interference with the ultrasound beam during echocardiographic examination is not known and has not been studied. Similar to air in the lung but to a lesser degree, silicone breast implants appear to prevent penetration of ultrasound beams. The poor penetration appears to be persistent and unrevealing despite increase in gain or change in the ultrasound wave's frequency.

Many women elect breast augmentation for cosmetic reasons. Women with congenital heart disease who have undergone cardiac surgery may have breast asymmetry or distortion and desire augmentation accordingly.

Knowledge of the extent of impairment of breast implants to the echocardiographic examination is important for few reasons:

1. Women with heart disease who need echocardiographic follow up and wish to undergo breast augmentation should be consulted as to the limitation of the echocardiographic examination following the procedure.
2. Women without heart disease considering breast augmentation should be informed of potential echocardiographic interference, if echocardiography be needed in the future,
3. Different surgical techniques may cause different masking effect.
4. Different implants size and shape may cause different masking effect.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Women with heart disease who need echocardiographic follow up and wish to undergo breast augmentation

Exclusion Criteria:

1. Unwillingness to participate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing breast augmentation
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion of women in which the breast implant will affect the quality of the Echo test. | one month
  The women will be gone through two Echo tests, the first before the operation and the second six weeks after the operation. The physician will compare the two tests.